CLINICAL TRIAL: NCT06136819
Title: Safety and Feasibility Dose Escalation Study for Evaluation of RT-310 for Treatment of Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostatic Hyperplasia (BPH)
Brief Title: RT-310 Dose Escalation BPH Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Resurge Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P18001
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: BPH (Benign Prostatic Hyperplasia); Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RT-310 Cohort 1 (Experimental): Combination Product: RT-310 implant Cohort 1
  Interventions: Combination Product: RT-310
- RT-310 Cohort 2 (Experimental): Combination Product: RT-310 Implant Cohort 2
  Interventions: Combination Product: RT-310

INTERVENTIONS:
Combination Product: RT-310 — Combination Product: RT-310 Implant for Investigational Treatment of Lower Urinary Tract Symptoms Secondary to BPH (Benign Prostatic Hyperplasia)

SUMMARY:
RT-310, a novel implant, is intended to minimally invasive treat locally the prostate gland for the management of prostate disease, while minimizing side-effects. The objectives of the study are to assess whether RT-310 is safe and feasible for the participant population.

DETAILED DESCRIPTION:
The RT-310 study is a first in human Phase 1 multi-center prospective, non-randomized dose escalation study to evaluate the safety and feasibility of RT-310 for treatment of Benign Prostatic Hyperplasia (BPH). Study participants will have placement of RT-310 and be followed through 180 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Male gender
* Diagnosis of symptomatic BPH
* Age ≥ 50 years up to 80 years
* International Prostate Symptom Score (IPSS) ≥ 13
* Prostate volume 30 to 80 cc per ultrasound
* Inadequate response and/or refusal of medical therapy for LUTS

Key Exclusion Criteria:

* Current urinary retention or at significant risk of urinary retention after drug washout
* Have an obstructive or protruding median lobe of the prostate
* Previous BPH surgical procedure or implants, urethral stricture, Any prior minimally invasive intervention (e.g. TUNA, Balloon, Microwave, Rezūm, UroLift) or surgical intervention of the prostate
* Previous pelvic surgery or irradiation
* History of neurogenic or atonic bladder
* Stress urinary incontinence, mixed or urge incontinence
* History of prostate or bladder cancer, confirmed or suspected malignancy of prostate or bladder
* History of compromised renal function or upper urinary tract disease
* Other co-morbidities that could impact the study results such as: severe cardiac arrhythmias uncontrolled by medications or pacemaker; congestive heart failure New York Heart Association (NYHA) III or IV; History of uncontrolled diabetes mellitus; significant respiratory disease in which hospitalization may be required
* Known immunosuppression (i.e. AIDS, post-transplant, undergoing chemotherapy)
* No more than two documented active urinary tract infections (UTI) by culture or bacterial prostatitis within last year documented by culture (UTI is defined as >100,000 colonies per ml urine from midstream clean catch or catheterization specimen)
* Current gross hematuria and/or visible hematuria with participant urine sample without known contributing factor
* Presence of a penile implant or stent(s) in the urethra or prostate
* PSA > 10 ng/ml unless prostate cancer is ruled out by biopsy. If PSA is > 4 ng/ml and ≤ 10 ng/ml, prostate cancer must be ruled out to the satisfaction of the investigator via additional tests including digital rectal exam (DRE) and/or biopsy
* Sensitivity to RT-310
* Unable to undergo magnetic resonance imaging (MRI) such as presence of cardiac pacemaker or implanted cardiac defibrillator
* Parkinson's disease or other neurologic disease that may impact bladder function such as stroke, TIA, multiple sclerosis

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Absence of unanticipated adverse events (UAEs) not listed in the protocol or Adverse Events (AEs) that meet the protocol definition of Serious Adverse Events (SAEs) | Baseline to Day 180
  Adverse events

SECONDARY OUTCOMES:
Change in prostate volume | Baseline to Day 180
  Transrectal ultrasound
Change in IPSS | Baseline to Day 180
  International Prostate Symptom Score (IPSS); IPSS scores range from 0 (no symptoms) to 35 (severe symptoms)
Uroflowmetry measure of Qmax | Baseline to Day 180
  Uroflowmetry measure of peak flow rate Qmax (mL/s)
Uroflowmetry measure of Qave | Baseline to Day 180
  Uroflowmetry measure of average flow rate, Qave (mL/s)
Uroflowmetry measure of voided volume | Baseline to Day 180
  Uroflowmetry measure of voided volume (mL)
PVR | Baseline to Day 180
  Post void residual (PVR) measurement

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Australian Clinical Trials, Wahroonga, New South Wales
  - Goldfields Urology, Bendigo, Victoria
  - Western Urology, Maribyrnong, Victoria
- Tauranga Urology Research, Tauranga, North Island, New Zealand